CLINICAL TRIAL: NCT04486976
Title: Comparative Study of the Cornea/Anterior Segment OCT CASIA2 and the RTVue XR OCT Avanti With AngioVue Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomey Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: TomeyCASIA2-001
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Glaucoma; Cataract
MeSH Terms: conditions — Glaucoma; Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Normal (Experimental)
  Interventions: Device: Cornea/Anterior Segment OCT CASIA2; Device: Optovue RTVue XR Avanti
- Glaucoma (Experimental)
  Interventions: Device: Cornea/Anterior Segment OCT CASIA2; Device: Optovue RTVue XR Avanti
- Cataract (Experimental)
  Interventions: Device: Cornea/Anterior Segment OCT CASIA2; Device: Optovue RTVue XR Avanti

INTERVENTIONS:
Device: Cornea/Anterior Segment OCT CASIA2 — Cornea/Anterior Segment OCT CASIA2 The Tomey Cornea/Anterior Segment OCT CASIA2 is a non-contact, high resolution tomographic and biomicroscopic device indicated for the in vivo imaging and measurement of ocular structures in the anterior segment, such as corneal thickness. The Tomey Cornea/Anterior Segment OCT CASIA2 is indicated as an aid in the visualization of anterior segment findings.
Device: Optovue RTVue XR Avanti — Optovue RTVue XR Avanti The Avanti is an optical coherence tomography system indicated for the in vivo imaging,axial cross-sectional, and three-dimensional imaging and measurement of anterior and posterior ocular structures.

SUMMARY:
This study is a prospective comparative, randomized, single center study to gather agreement and precision data in all subjects.

ELIGIBILITY:
Inclusion Criteria - Normal Group:

1. Male or female subjects 22 years of age or older who have full legal capacity to volunteer on the date the informed consent is signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date;
3. Subjects who agree to participate in the study;

Exclusion Criteria - Normal Group:

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects with any current ocular pathology, as determined by self-report and confirmed by the investigator assessment and/or confirmed by the investigator assessment at the study visit;
3. Subjects that present with an active ocular infection in either eye;
4. Subjects who have a history of ocular surgery, including laser therapy/surgery;
5. Subjects with a condition or in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Inclusion Criteria - Cataract Group:

1. Male or female subjects 22 years of age or older who have full legal capacity to volunteer on the date the informed consent is signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date;
3. Subjects who agree to participate in the study;
4. Subjects diagnosed with cataract classified per the LOCS III scale;

Exclusion Criteria - Cataract Group:

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects with corneal or conjunctival abnormalities that may affect adequate assessment of the anterior chamber in either eye;
3. Subjects that present with an active ocular infection in either eye;
4. Subjects who have a history of ocular surgery, including laser therapy/surgery;
5. Subjects with a condition or in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Inclusion Criteria - Glaucoma Group:

1. Male or female subjects 22 years of age or older who have full legal capacity to volunteer on the date the informed consent is signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date;
3. Subjects who agree to participate in the study;
4. Subjects with glaucomatous optic nerve damage as evidenced by any of the following optic disc or retinal nerve fiber layer structural abnormalities:

   1. Diffuse thinning, focal narrowing, or notching of the neuroretinal rim, especially at the inferior or superior poles with or without disc hemorrhage;
   2. Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue
5. History of Visual field defects within the previous six (6) months from the study visit or measured the day of the study visit consistent with glaucomatous optic nerve damage with at least one of the following two findings:

   1. On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level;
   2. Glaucoma hemi-field test "outside normal limits."

Exclusion Criteria - Glaucoma Group:

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects with corneal or conjunctival abnormalities that may affect adequate assessment of the anterior chamber in either eye;
3. Subjects that present with an active ocular infection in either eye;
4. No reliable Humphrey Field Analyzer (HFA) visual field (24-2 Sita Standard, white on white) result within 6 months of the study visit, defined as fixation losses > 33% or false positives > 33%, or false negatives > 33% in the study eye;
5. Subjects with a condition or in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2020-06-27 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Agreement of Corneal thickness (μm) measurement for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT | Up to 30 days
  Thickness of Cornea
Agreement of Angle-Opening Distance (mm) measurement for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT | Up to 30 days
  Angle-Opening Distance Angle-Opening Distance
Agreement of Trabecular-Iris Space Area measurement (mm²) for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT | Up to 30 days
  Trabecular-Iris Space Area
Agreement of OCT image quality for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT and evaluation of visibility of predefined anatomical structures | Up to 30 days
Precision of the Corneal thickness (μm) measurement for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT | Up to 30 days
  Corneal thickness
Precision of the Angle-Opening Distance (mm) measurement for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT | Up to 30 days
  Angle-Opening Distance
Precision of the Trabecular-Iris Space Area measurement (mm²) for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT | Up to 30 days
  Trabecular-Iris Space Area
Precision of the Anterior Corneal Depth measurement (mm) for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT | Up to 30 days
  Anterior Corneal Depth
Precision of the Anterior Corneal Width measurement (mm) for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT | Up to 30 days
  Anterior Corneal Width
Precision of the Pupil Diameter measurement (mm) for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT | Up to 30 days
  Pupil Diameter
Precision of the Ks (steep meridian) measurement (D) for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT | Up to 30 days
  Ks (steep meridian)
Precision of the Kf (flat meridian) measurement (D) for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT | Up to 30 days
  Kf (flat meridian)
Precision of the Corneal Cylinder measurement (D) for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT | Up to 30 days
  Corneal Cylinder
Precision of the Average Keratometry measurement (D) for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT | Up to 30 days
  Average Keratometry
Precision of the Angle Recess Area measurement (mm²) for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT | Up to 30 days
  Angle Recess Area
Precision of the Trabecular-Iris Angle measurement (mm) for Cornea/Anterior Segment OCT CASIA2 and Optovue RTVue XR Avanti OCT | Up to 30 days
  Trabecular-Iris Angle

SECONDARY OUTCOMES:
Adverse Events | Up to 30 days
  An adverse event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational device but not necessarily related to the investigational device.

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No